CLINICAL TRIAL: NCT05332236
Title: Validierung Eines Psychometrischen Fragebogens Zur Eltern-Kind-Kommunikation im Selbstbericht
Brief Title: Parent-adolescent Communication: Validation of a German Language Scale and Its Longitudinal Association With Adolescent Mental Health
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: E-K-Kom-Val
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Parent-Child Relations
Keywords: parent-child communication, parent-adolescent communication

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Community sample: Adolescents (10-18 years) and their parents, recruited via online sampling, from the general population
  Interventions: Diagnostic Test: Parent-Adolescent Communication Scale (questionnaire)
- At-risk sample: Parents seeking parenting advice in information centres/helplines.
  Interventions: Diagnostic Test: Parent-Adolescent Communication Scale (questionnaire)
- Clinical sample: Children and parents are recruited among in- and outpatients at the Clinic for Child and Adolescent Psychiatry of the University Medical Center Hamburg-Eppendorf
  Interventions: Diagnostic Test: Parent-Adolescent Communication Scale (questionnaire)

INTERVENTIONS:
Diagnostic Test: Parent-Adolescent Communication Scale (questionnaire) — Observational psychometric validation study

SUMMARY:
A German version of the Parent-Adolescent Communication Scale (PACS, Barnes & Olson, 1982) will be validated in a large sample of children (10-18 years) and their parents. As a secondary objective, the association of communication quality, children's somatic symptoms and mental health will be explored. After two years, participants from the community sample will be contacted again to see whether baseline communication quality predicts adolescent mental health two years later.

DETAILED DESCRIPTION:
The quality of parent-child communication (pcc) is likely to be of importance for child mental health, especially during adolescence. Therefore, pcc is relevant in etiologic research, diagnostics, and as a possible target for intervention in at-risk and clinical populations.

Up to now, there is no validated questionnaire in German language to assess pcc as parent and child self-report. A German translation of the widely used Parent-Adolescent Communication Scale (PACS, Barnes & Olson, 1982) will be validated in this study. This questionnaire comprises 20 items that are identical in parent and child versions apart from the referent (my mother/my father/my daughter/my son). In the original scale, two subscales were found via factor analysis: Open communication and problems in communication (ten items each). Internal consistency was adequate in most studies. Several studies have shown associations between pcc and child mental health.

In the current study, the primary aim is to validate the questionnaire in a community, an at-risk, and a clinical sample, with the at-risk sample comprising parent-child dyads with parents seeking parenting advice. The clinical sample will be recruited among in- and outpatients at the Clinic for Child and Adolescent Psychiatry of the University Medical Center Hamburg-Eppendorf. Discriminative validity will be assessed in terms of group differences, construct validity in terms of correlations with different subscales on the parent-child relationship. With regard to the factorial structure, an exploratory factor analysis will be performed. As a secondary aim, the association between somatic symptoms, mental health, and pcc will be studied.

In the longitudinal part of the study, parent-child communication quality will be analysed as a predictor of mental health, especially depressive symptoms and somatic symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate
* Child age: 10-18 years.

Exclusion Criteria:

- None.

Ages: 10 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children and their parents from the general population, parents seeking advice in parenting support centres and their children, parents and children recruited among in- and outpatients at the Clinic for Child and Adolescent Psychiatry of the University Medical Center Hamburg-Eppendorf
Sampling Method: Probability Sample
Enrollment: 2338 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Parent-adolescent communication scale | Baseline
  20 item measure consisting of two subscales (open and problem communication), 5-point Likert scale; child and parent report
Change in general adolescent mental health | From baseline to 2 years after recruitment
  Changes in general adolescent mental health will be measured with the Strengths and Difficulties Questionnaire (SDQ), total scale. The total scale consists of 20 items rated on a 3-step scale. Higher values indicate higher symptom burden.

SECONDARY OUTCOMES:
Depressive symptoms two years after recruitment | Two years after initial recruitment.
  The Centre for Epidemiological Studies Depression Scale for Children (DES-DC) measures depressive symptoms in adolescents using 20 items on a four-step Likert scale. Higher values indicate higher symptom burden. Instead of general cut-offs, standardized T-values accoring to gender groups above 60 can be considered as conspicuous (Barkmann et al. 2011).
Change in somatic complaints | From baseline to two years after recruitment.
  The somatic complaints subscale of the Child Behavior Checklist/Youth Self Report questionnaire will be used to measure somatic complaints in adolescents. It consists of 7 items and is measured on a three-step Likert scale. Higher values indicate more and more frequent somatic complaints.

CONTACTS AND LOCATIONS:
Overall Officials: Holger Zapf, PhD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zapf H, Boettcher J. Psychometric evaluation of the german version of the parent-adolescent communication scale. Eur Child Adolesc Psychiatry. 2025 Mar;34(3):1097-1109. doi: 10.1007/s00787-024-02541-4. Epub 2024 Aug 7. PMID 39110191
- [Derived] Zapf H. Parent-adolescent communication quality does not moderate the association of emotional burden and somatic complaints in adolescents: a cross-sectional structural equation model. Child Adolesc Psychiatry Ment Health. 2025 Mar 22;19(1):28. doi: 10.1186/s13034-025-00882-9. PMID 40121474